CLINICAL TRIAL: NCT03947476
Title: Extrapulmonary Lung Protection Strategy for Patients With Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EXPECT
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-05

CONDITIONS: Mechanical Ventilation; Ventilator-induced Lung Injury; Transpulmonary Pressure
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: thoracic band — Thoracic band fixation

SUMMARY:
As an important life sustaining support , mechanical ventilation has greatly promoted the development of modern intensive care units. However, mechanical ventilation can lead to ventilator-induced lung injury, including barotrauma, volutrauma, atelectrauma and biotrauma. All patients undergoing mechanical ventilation are at risk of barotrauma. A multicenter prospective cohort study of 5183 patients with mechanical ventilation showed that the incidence of pulmonary barotrauma was 3%. The incidence of pulmonary barotrauma varied according to the causes of mechanical ventilation: chronic obstructive pulmonary disease (3%), asthma (6%), chronic interstitial lung disease (10%), acute respiratory distress syndrome (7%) and pneumonia (4%).

At present, it is considered that one of the main causes of barotrauma is the increasing of transpulmonary pressure. Transpulmonary pressure is the difference between alveolar pressure and intrapleural pressure. The commonly adopted lung protective ventilation methods include: limiting plateau pressure less than or equal to 30 cmH2O, using small tidal volume ventilation (6-8 mL/kg ideal body weight) . All the above methods are to reduce trans-pulmonary pressure by reducing alveolar pressure. In addition to reducing alveolar pressure, increasing pleural pressure is another important way to reduce transpulmonary pressure and the incidence of barotrauma. At present, the main method is the use of neuromuscular blockade. However, there are many shortcomings in of neuromuscular blockade: 1. Time limit, generally not more than 48 hours; 2. Long-term use of neuromuscular blockade causes adverse reactions such as myopathy; 3. Neuromuscular blockade are only suitable for invasive mechanical ventilation patients, but not for non-invasive mechanical ventilation or high flow oxygen inhalation patients. Therefore, it is urgent to find other methods to reduce trans-pulmonary pressure and lung injury.

The investigators drew inspiration from the early mechanism of "iron lung" ventilator and the clinical practice of reducing trans-pulmonary pressure and lung injury in obese patients. In the early stage, the investigators carried out the clinical practice of extrapulmonary lung protection strategy, that is, to give thoracic band restraint to patients undergoing non-invasive mechanical ventilation so as to reduce chest wall compliance, which can be significantly reduced under the same inspiratory pressure and occurrence of barotrauma. However, the respiratory mechanics mechanism of this method still needs to be further studied to determine whether it can reduce the incidence of barotrauma by reducing transpulmonary pressure. It is accessible and inexpensive. The aim of this study was to determine the changes of transpulmonary pressure in patients with invasive mechanical ventilation before and after thoracic band fixation by esophageal manometry without spontaneous breathing.

ELIGIBILITY:
Inclusion Criteria:

1. BMI > 18, BMI < 40
2. Age > 18 years old
3. Patients who need invasive mechanical ventilation for lower abdominal surgery, brain surgery, cerebral hemorrhage and cerebral infarction
4. Mechanical ventilation at least 12 hours

Exclusion Criteria:

1. BMI < 18 or BMI > 40
2. Age < 18 years old
3. abstain from nasogastric tube
4. Pneumothorax
5. Pregnant women
6. Patients with severe hypoxemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit who need invasive mechanical ventilation at least 12 hours
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Inspiratory of transpulmonary pressure | up to 24 hours
  Measurement of transpulmonary pressure by placement of esophageal manometer tube during inspiratory,the metric is cmH2O
Expiratory of transpulmonary pressure | up to 24 hours
  Measurement of transpulmonary pressure by placement of esophageal manometer tube during expiratory,the metric is cmH2O

CONTACTS AND LOCATIONS:
Overall Officials: Minjie Ju, PHD, Principal Investigator — Fudan University
Locations (1):
- Ju Minjie, Shanghai, Shanghai Municipality, China